CLINICAL TRIAL: NCT04637048
Title: Observational Study on Patients With Hepatobiliary Tumors
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Gang Chen, MD (Other)
Responsible Party: Sponsor-Investigator, Gang Chen, MD, Division Chief of Education; Deputy Director of Hepatobiliary Surgery, First Affiliated Hospital of Wenzhou Medical University
Organization: First Affiliated Hospital of Wenzhou Medical University (Other)
Other Study IDs: Obs-Hepatobiliary CA
Record Dates: First submitted 2020-11-14; First posted 2020-11-19 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Hepatocellular Carcinoma; Cholangiocarcinoma; Gallbladder Cancer; Biliary Tract Cancer; Gastric Cancer; Colorectal Cancer
Keywords: Hepatocellular Carcinoma; Cholangiocarcinoma; Gallbladder Cancer; Biliary Tract Cancer; blood sample; tissue sample; stool sample
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma; Gallbladder Neoplasms; Biliary Tract Neoplasms; Stomach Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — normal tissue, tumor samples, blood, urine, feces, ascites, bile samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hepatobiliary tumors have a poor prognosis and high individual heterogeneity, the patient with hepatobiliary tumors even accepted radical surgery, the postoperative recurrence rate is still high. Therefore, it is of great significance to find important prognostic markers to improve patient prognosis and formulate new treatment plans. In recent years, targeted therapy and immunotherapy make cancer treatment enter a new field, However, tumor heterogeneity is the greatest challenge in cancer therapeutics and biomarkers discovery. In this study, we collected a wide rang of patients' information, including photos of patients' face, physical strength and nutrition indicators, blood ,stool and pathological tissue specimens from tumor patients, then Multi-omics testing were applied to Looking for novel therapeutic targets and prognostic markers to predict patient response to treatment. Clinicians choose the best treatment plan for the patient based on the test results to improve the patient's survival time and quality of life.

DETAILED DESCRIPTION:
This is an ongoing, longitudinal, observational clinical cohort study of patients with tumors of the alimentary tract, mainly hepatobiliary tumors. All the patients are diagnosed, treated and followed up. In the future, some other patient information will be gradually updated to this database

ELIGIBILITY:
Inclusion Criteria:

1. Be older than 18 years old;
2. Clinical or pathological diagnosis of malignant hepatobiliary tumors;
3. Patients have received or are about to receive surgery, chemotherapy radiotherapy, targeted therapy, local therapy, immunotherapy, etc;
4. Patients understand and are willing to sign written informed consent.

Exclusion Criteria:

1. Patients considered by the doctor to be unsuitable for entry into this study (mental disorder or poor compliance, etc.);
2. The patient or guardian is unwilling to participate in this study;
3. Pregnant women;
4. Combined with other serious systemic diseases (heart failure, renal failure,hematopoietic system disease or Uncontrollable acute infection);
5. Estimated survival time is less than 1 month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed and treated as hepatobiliary tumors and other alimentary tract tumors
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-02-16 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the overall survival rate of all patients with hepatobiliary tumor | 5 years
  In order to identify the potential influence factors of hepatobiliary tumor patients survival

SECONDARY OUTCOMES:
Evaluate the recurrence free survival rate of patients with hepatobiliary tumor | 5 years
  In order to identify the potential influence factors of tumor recurrencesamples from patients with hepatobiliary cancers
Evaluate the cancer-specific survival rate of patients with hepatobiliary tumor | 5 years
  In order to identify the potential influence factors of tumor-induced death in patients with hepatobiliary tumors
Evaluate the Progression Free Survival rate of patients with hepatobiliary tumor | 5 years
  In order to identify the potential influence factors of tumor progression from patients with hepatobiliary cancers

CONTACTS AND LOCATIONS:
Overall Officials: Gang Chen, M.D., Principal Investigator — First Affiliated Hospital of Wenzhou Medical University
Locations (1):
- Gang Chen, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang J, Wang D, Ma L, An X, Hu Z, Zhu H, Zhang W, Chen K, Ma J, Yang Y, Wu L, Chen G, Wang Y. Sarcopenia negatively affects postoperative short-term outcomes of patients with non-cirrhosis liver cancer. BMC Cancer. 2023 Mar 6;23(1):212. doi: 10.1186/s12885-023-10643-6. PMID 36879265